CLINICAL TRIAL: NCT01489306
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Inhaled MDT-637 Administered to Healthy Volunteers for 10 Days
Brief Title: A Trial to Assess the Safety, Tolerability and Pharmacokinetics of MDT-637 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MicroDose Therapeutx, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDT-637-CP-102
Record Dates: First submitted 2011-12-07; First posted 2011-12-09 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Drug Safety
Keywords: Respiratory Syncytial Virus Infection; RSV
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — VP-14637

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- MDT-637 (Experimental): Active formulation
  Interventions: Drug: MDT-637
- Placebo (Placebo Comparator): Matched Placebo Comparator
  Interventions: Drug: MDT-637

INTERVENTIONS:
Drug: MDT-637 — Inhaled doses of MDT-637 over a 10 day period
  Arms: MDT-637
Drug: MDT-637 — Inhaled doses of MDT-637 over a 10 day period
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the tolerability and safety of a range of repeated inhaled doses of MDT-637. This includes monitoring effects on pulmonary function and determination of blood levels of MDT-637 following inhalation.

ELIGIBILITY:
Inclusion Criteria:

* Males and/or surgically sterile or post-menopausal females (confirmed by FSH test); males must agree to practice barrier contraception until they are discharged from the study
* Willing to give written informed consent
* 18 to 50 years of age
* BMI of 19-30 kg/m2
* Non-smoker (for at least 90 days prior to screening) and willing to abstain from smoking during the course of the study
* Good general health as determined by medical history, physical examination, spirometry, ECG and clinical laboratory tests
* Willing to abstain from alcohol, caffeine, and xanthine-containing beverages for 24 hours prior to and 24 hours after dosing

Exclusion Criteria:

* Uncontrolled, clinically significant disease which in the opinion of the Principal Investigator and Sponsor (MDTx) would place the subject at risk through study participation or would confound the assessment of the safety of MDT-637
* Evidence of current or history of respiratory disease; for instance asthma, emphysema, chronic bronchitis or cystic fibrosis.
* Upper respiratory tract infection within 6 weeks of Visit 1
* Symptoms of rhinitis (stuffy nose, rhinorrhea, sneezing, nasal discharge) within 2 weeks of Visit 1
* Current symptoms of cough, dyspnea, wheezing or nocturnal awakenings due to respiratory symptoms
* History of significant nasal irritation from nasal inhalation of medication
* History of malignancy
* History of clinically significant alcohol or drug abuse
* Positive drug screen for drugs of abuse
* Positive test for HIV, Hepatitis B or Hepatitis C
* Allergy to lactose, or lactose intolerance
* Use of prescription medication within 14 days of Visit 2 or over-the-counter preparations, including dietary and herbal supplements, within 5 days of Visit 2
* Positive urine pregnancy test at Visit 1
* Inability to perform reproducible spirometry in accordance with American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines
* Abnormal QTc interval at Visit 1(>450 msec in males or > 470 msec in females)
* Significant blood donation (or testing) in previous 8 weeks

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of 3 escalating doses of MDT-637 dry powder inhalation in healthy volunteers | Up to 48 days (including up to 28 days of screening period)
  Safety measurements include Clinical Laboratory Evaluations, Pulmonary Function Tests (Spirometry), ECG, Vital Signs, Physical Examination and Assessment of Adverse Events.

SECONDARY OUTCOMES:
Plasma pharmacokinetics for MDT-637 dry powder inhalation | Multiple plasma samples collected during the dosing period, upto 24 hr post last dose
  Plasma Samples will be measured to determine MDT-637 pharmacokinetics

CONTACTS AND LOCATIONS:
Locations (1):
- West Coast Clinical Trials, Cypress, California, United States

REFERENCES:
- See also: Related Info — http://mdtx.com/pipeline/proprietary-products/mdt-637/